CLINICAL TRIAL: NCT06122233
Title: A Randomised Clinical Trial of a Digital Self-management Package for People With Interstitial Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Monash University (Other); Lung Foundation Australia (Unknown); University of Tasmania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: X23-0387
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Lung Diseases, Interstitial; Pulmonary Fibrosis
Keywords: Self-Management; Chronic diseases
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, blinding will not be possible for participants and care providers (i.e. healthcare professionals making phone calls to participants). Where practicable, members of the investigative team will be blinded. Outcome assessors will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REBUILD-SM Group (Experimental): Participants randomised to the intervention will receive the self-management package, including the REBUILD app. Structured self-management support via telephone or Zoom call will be provided 4 times during the 12-week intervention period.
  Interventions: Behavioral: Pulmonary Fibrosis self-management package and smartphone application
- Standard Care Group (No Intervention): In the control arm, participants will receive standard care and a reduced capability version of the REBUILD app to be used for data-capture only. They will also receive phone/Zoom calls at the same frequency during the 12-week intervention period, but no health advice will be given. After 26 weeks, participants in this group will receive access to the fully functional REBUILD app, however they will not receive the self-management content or the support phone calls provided to the intervention group.

INTERVENTIONS:
Behavioral: Pulmonary Fibrosis self-management package and smartphone application — The pulmonary fibrosis package includes modules on understanding treatment options for pulmonary fibrosis, managing medication and side effects, understanding and accessing clinical trials, managing shortness of breath, managing fatigue and mood, managing co-existing conditions, the role and importance of pulmonary rehabilitation and regular physical activity, role of oxygen therapy, smoking cessation advice and support, accessing community support, and communicating with others when living with pulmonary fibrosis.
  The RE-BUILD app is used as a tool for data collection and to help participants self-monitor their disease over time. Participants enter their health data, including baseline conditions, medications and diagnosis, pulmonary function results and supplementary oxygen use. It also tracks air quality data close to the participant as well as physical activity level (step count). The app also has links to ILD-related educational resources.
  Other Names: REBUILD-SM
  Arms: REBUILD-SM Group

SUMMARY:
The goal of this clinical trial is to compare REBUILD-SM (a purpose-built smartphone app and self-management package) with standard care in people with interstitial lung disease (ILD). The main question it aims to answer is:

• Does REBUILD-SM improve health-related quality of life, symptoms, anxiety, self-efficacy and physical activity for people with ILD?

Participants in the intervention group will work through the self-management package with support from a healthcare professional via phone or Zoom. They will also enter deidentified health data into the RE-BUILD smartphone app to track their progress over time. Participants in the control group will use a reduced functionality version of the smartphone app only.

Researchers will compare both groups to see if there is any difference in health-related quality of life, symptoms, anxiety, self-efficacy and level of physical activity.

DETAILED DESCRIPTION:
This study compares REBUILD-SM with standard care in people with ILD. REBUILD-SM comprises a purpose-built smartphone app that allows subjects to enter and track health data over time and an integrated self-management package.

Participants will enter their respiratory diagnosis, medications and side effects, weight, lung function test results, oxygen saturation level and supplemental oxygen usage into the smartphone app. They will also complete questionnaires at specific timepoints using the app. Participants will input most of this data at the beginning of the trial and update it when it changes, for example, after obtaining a new lung function result, starting a new medication, or getting a new side effect from an existing medication. Entering data into the app is expected to take around 30 minutes at the start of the trial, and about 20 minutes at 12, 26 and 52 weeks when completing the questionnaires. Updating data is expected to take about 5-10 minutes and will only happen when there is a change, for example, once per week, although it may not be this frequent.

The app will not provide any recommendations on the health data participants enter - it is simply for recording purposes. To ensure data collection is as complete as possible, electronic reminders will be sent to participants when questionnaires are not completed at the specified timepoints and will alert the study team if the participant fails to complete the questionnaires after the reminder. This will prompt a phone call from a member of the study team to encourage the participant to complete the endpoints. App analytics will be used in the data analysis phase (after the trial is over) to understand how participants have engaged with the app.

Participants in the intervention group will be asked to log into and use the self-management website or view the content via the REBUILD app with support from the study team. The self-management content includes 13 modules and has been designed in collaboration with people with ILD to help increase their ability to self-manage their chronic disease.

During the intervention period, participants will receive four phone calls from a health professional involved in the management of people with ILD to help them set health-related goals and identify appropriate modules from the website to help achieve these goals. These four phone calls are expected to take about 15-30 minutes each.

Each module provides information regarding the topic and provides access to relevant websites, fact sheets, booklets, videos and webinars as well as other external resources. Participants will have direct access to these external resources from within the package through hyperlinks embedded in the title of each resource. Participants are expected to work through their selected modules at their own pace - there is no specific amount of time they are required to allocate to the intervention, and they can utilize as many or as few of the resources as they like.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibrotic ILD
* In possession of a smartphone/tablet and an email address
* Able to understand written and spoken English
* Adequate digital literacy to complete requirements of trial
* On stable ILD treatment for 30 days prior to enrolment

Exclusion Criteria:

* Not in possession of a smartphone/tablet
* Insufficient digital literacy to complete requirements of trial
* Unable to communicate in written/spoken English
* Not on stable ILD treatment for 30 days prior to enrolment
* Acute exacerbation within 30 days prior to enrolment
* Participating in pulmonary rehab at enrolment or during 12-week intervention period
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in King's Brief Interstitial Lung Disease (K-BILD) questionnaire score | Baseline and 12 weeks post-randomisation
  Score range 0 - 100; higher score corresponding to better outcome.

SECONDARY OUTCOMES:
Change in K-BILD score | 26 and 52 weeks post-randomisation
  As above
Change in European Quality of Life 5-Dimensions 5-Level (EQ-5D-5L) questionnaire score | Baseline, 12, 26 and 52 weeks post-randomisation
  Score range 11111 - 55555; 0-100; higher score indicating worse outcome
Change in General Self-Efficacy Scale score | Baseline, 12, 26, and 52 weeks post-randomisation
  Score range 10 - 40; higher score indicating low level of perceived self-efficacy
Change in Dyspnoea-12 score | Baseline, 12, 26 and 52 weeks post-randomisation
  Score range 0-36; higher score corresponding to greater level of dyspnoea
Change in Hospital Anxiety and Depression Scale score | Baseline, 12, 26 and 52 weeks post-randomisation
  Score range 0-21 (for anxiety and depression); higher scores corresponding to severe anxiety and/or depression
Change in physical activity levels | Baseline, 12 and 52 weeks post-randomisation
  Change in steps per day and change in time spent in the four intensity categories (inactive, low, medium and high activity) will be measured using a physical activity monitor
Uptake/ changes to ILD treatments | Baseline, 12, 26 and 52 weeks post-randomisation
  Includes changes to medications, commencement or change in supplemental oxygen use, participation in pulmonary rehab
Change in mHealth App Usability questionnaire (MAUQ) score | 12, 26 and 52 weeks post-randomisation
  Score range 18-126; higher score indicating greater satisfaction with the REBUILD app
Change in e-Health Literacy (eHEALS) questionnaire score | Baseline,12 and 52 weeks post-randomisation
  Score range 8-40; higher score indicating higher degree of perceived e-health literacy
Health Care Climate questionnaire | 12 weeks post-randomisation
  Score range 6-42; higher score indicating greater satisfaction with treating team

CONTACTS AND LOCATIONS:
Overall Officials: Tamera Corte, Principal Investigator — University of Sydney; Dan Chambers, Principal Investigator — The University of Queensland; Nicole Goh, Principal Investigator — Institute of Breathing and Sleep; Ian Glaspole, Principal Investigator — The Alfred
Locations (4):
- Australia (4):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Alfred Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be placed in a secure repository for future analysis.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available at the end of the trial (approx. April 2028).
Access Criteria: Requires ethical approval

REFERENCES:
- [Derived] Barton C, Hoffman M, Cox NS, Glenn LM, Lee JYT, Cox I, Goh NSL, Troy LK, Mackintosh J, Chambers DC, Glaspole IN, Gebski V, Keech A, Palmer A, Laranjo L, Knibbs LD, Moodley Y, Brooke M, Holland AE, Corte TJ. A randomised clinical trial of a digital self-management package for people with interstitial lung disease: the REBUILD-SM protocol. Respir Res. 2025 Dec 5;27(1):14. doi: 10.1186/s12931-025-03442-z. PMID 41350860